CLINICAL TRIAL: NCT00945061
Title: Partial Breast Re-Irradiation for Patients With Ipsilateral Breast Tumor Recurrence, After First Being Treated With Breast Conservation for Early Stage Breast Cancer: An Efficacy Trial Comparing Mammosite® and Intraoperative Radiation
Brief Title: Radiation Therapy in Treating Patients With Recurrent Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE11107
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; recurrent breast cancer; invasive ductal breast carcinoma; medullary ductal breast carcinoma with lymphocytic infiltrate; mucinous ductal breast carcinoma; papillary ductal breast carcinoma; tubular ductal breast carcinoma; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Breast Neoplasms, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intraoperative radiation therapy (Experimental): Patients undergo partial breast irradiation delivered as a single intra-operative radiation dose to the tumor bed.
  Interventions: Radiation: intraoperative radiation therapy
- Intracavitary balloon brachytherapy (Experimental): Patients undergo partial breast irradiation delivered as MammoSite® brachytherapy consisting of 10 fractions over 5 days.
  Interventions: Radiation: intracavitary balloon brachytherapy

INTERVENTIONS:
Radiation: intracavitary balloon brachytherapy — Patients undergo brachytherapy
  Arms: Intracavitary balloon brachytherapy
Radiation: intraoperative radiation therapy — Patients undergo radiotherapy
  Arms: Intraoperative radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. It is not yet known whether a single dose of radiation therapy is more effective than implant radiation therapy for 5 days in treating patients with recurrent breast cancer.

PURPOSE: This phase II trial is studying implant radiation therapy to see how well it works compared with radiation therapy during surgery in treating patients with recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the in breast recurrence rate following repeat radiation to the breast. These patients will be followed for a period of five years following completion of radiation to determine these rates.
* To determine the cosmetic outcome resulting from partial breast re-irradiation using different techniques, including both physician and patient rated scales.
* To determine patient satisfaction of partial breast re-irradiation as it pertains to their overall treatment experience, as measured by a questionnaire.
* To determine if there are patient factors illuminated during a discussion of informed consent, which limit a patient's suitability to receive partial breast re-irradiation delivered by a particular technique.
* To evaluate tylectomy wound healing and overall complication rate after partial breast re-irradiation.
* To determine ipsilateral breast tumor recurrence rates and tumor bed recurrence rates.These patients will be followed for a period of five years following completion of the second course of radiation to determine these rates.

OUTLINE: Patients are stratified according to which modality is best suited for the patient. Patients are assigned to 1 of 2 groups.

All patients undergo excisional biopsy or needle localization removal of the tumor. Patients with margins < 2 mm undergo re-excision of the biopsy cavity.

* Group 1: Patients undergo partial breast irradiation delivered as a single intra-operative radiation dose to the tumor bed.
* Group 2: Patients undergo partial breast irradiation delivered by Mammosite® brachytherapy consisting of 10 fractions over 5 days.

Quality of life is assessed at baseline, 1 month after completion of radiotherapy, and then at follow-up visits.

After completion of study treatment, patients are followed up at 1 month, every 3 months for 1 year, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients' recurrences must have histologically confirmed ductal carcinoma in-situ, invasive ductal, medullary, papillary, colloid (mucinous), or tubular histologies.
* Lesion size ≤ 3 cm treated with a tylectomy and whole breast irradiation (with or without tumor bed boost)
* Unifocal breast cancer recurrence
* Negative resection margins with at least a 2 mm margin from invasive and in situ cancer or a negative re-excision
* Hormonal therapy is allowed. If chemotherapy is planned, the radiation is delivered first and chemotherapy must begin no earlier than two weeks following completion of radiation.
* Signed study-specific informed consent prior to study entry.

Exclusion Criteria:

* Patients with distant metastatic disease
* Patients with invasive lobular carcinoma, extensive lobular carcinoma in-situ, extensive ductal carcinoma in-situ (spanning more than 3 cm), or nonepithelial breast malignancies such as lymphoma or sarcoma.
* Patients with multicentric carcinoma (tumors in different quadrants of the breast or tumors separated by at least 4 cm). Palpable or radiographically suspicious contralateral axillary, ipsilateral or contralateral supraclavicular, infraclavicular, or internal mammary lymph nodes unless these are histologically or cytologically confirmed negative.
* Extensive intraductal component (EIC) by the Harvard definition, i.e. 1) more than 25% of the invasive tumor is Ductal carcinoma in situ (DCIS) and DCIS present in adjacent breast tissue. Presence of an EIC increases the chance of local recurrence, and as such, one might not be a candidate for repeat breast conservation.
* Patients with Paget's disease of the nipple.
* Patients with skin involvement.
* Patients with collagen vascular disorders, specifically systemic lupus erythematosis, scleroderma, or dermatomyositis.
* Patients with psychiatric, neurologic, or addictive disorders that would preclude obtaining informed consent.
* Other malignancy, except non-melanomatous skin cancer, < 5 years prior to participation in this study.
* Patients who are pregnant or lactating due to potential fetal exposure to radiation and unknown effects of radiation on lactating females.
* Patients with known BReast CAncer gene (BRCA)1/BRCA 2 mutations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-09-23 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Lyons, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Started | 12 | 1
Completed | 12 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy | Total
Number analyzed (Participants) | 12 | 1 | 13
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 1 | 0 | 1
  50-59 years | 4 | 0 | 4
  60-69 years | 4 | 1 | 5
  70-79 years | 1 | 0 | 1
  80-89 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 1 | 13
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 1 | 12
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 9 | 1 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: Percent of participants with Ipsilateral breast tumor recurrence (IBTR). IBTR includes: true recurrence (TR) thought to occur when residual cancer cells grow gradually to detectable size and new primary (NP) thought to be new cancer independently arising in the preserved breast.
Time Frame: 1 month after radiation therapy (RT)
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 12 | 1
percentage of participants | 0 | 0

2. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: as for outcome 1
Time Frame: 3 months after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 0 | 0

3. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: as for outcome 1
Time Frame: 6 months after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 0 | 0

4. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: as for outcome 1
Time Frame: 9 months after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 0 | 0

5. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: as for outcome 1
Time Frame: 12 months after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 0 | 0

6. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: as for outcome 1
Time Frame: 2 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

7. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: as for outcome 1
Time Frame: 3 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

8. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: as for outcome 1
Time Frame: 4 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 10 | 1
percentage of participants | 10 | 0

9. Primary Outcome: Ipsilateral Breast Tumor Recurrence Rates
Description: as for outcome 1
Time Frame: 5 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 9 | 1
percentage of participants | 11 | 0

10. Primary Outcome: Tumor Bed Recurrence Rates
Description: Percent of participants with tumor bed recurrence, defined as recurrence in the same quadrant as the surgical excision
Time Frame: 1 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 12 | 1
percentage of participants | 0 | 0

11. Primary Outcome: Tumor Bed Recurrence Rates
Description: Percent of participants with tumor bed recurrence, defined as recurrence in the same quadrant as the surgical excision
Time Frame: 3 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 0 | 0

12. Primary Outcome: Tumor Bed Recurrence Rates
Description: Percent of participants with tumor bed recurrence, defined as recurrence in the same quadrant as the surgical excision
Time Frame: 6 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 0 | 0

13. Primary Outcome: Tumor Bed Recurrence Rates
Description: Percent of participants with tumor bed recurrence, defined as recurrence in the same quadrant as the surgical excision
Time Frame: 12 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 0 | 0

14. Primary Outcome: Tumor Bed Recurrence Rates
Description: Percent of participants with tumor bed recurrence, defined as recurrence in the same quadrant as the surgical excision
Time Frame: 2 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

15. Primary Outcome: Tumor Bed Recurrence Rates
Description: Percent of participants with tumor bed recurrence, defined as recurrence in the same quadrant as the surgical excision
Time Frame: 3 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

16. Primary Outcome: Tumor Bed Recurrence Rates
Description: Percent of participants with tumor bed recurrence, defined as recurrence in the same quadrant as the surgical excision
Time Frame: 4 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 10 | 1
percentage of participants | 10 | 0

17. Primary Outcome: Tumor Bed Recurrence Rates
Description: Percent of participants with tumor bed recurrence, defined as recurrence in the same quadrant as the surgical excision
Time Frame: 5 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 9 | 1
percentage of participants | 11 | 0

18. Primary Outcome: Cosmetic Outcome as Determined by an Established Scale
Description: Cosmetic outcome as determined by four-level scale of cosmetic outcome scale, with levels poor, fair, good, and excellent in increasingly positive outcomes.
  Excellent: Minimal or no difference in the size or shape of the treated breast Good: Slight difference in the size or shape of the treated breast Fair: Obvious difference in the shape and size of the treated breast Poor: Obvious difference in the shape and size of the treated breast
Time Frame: 1 month after RT & Q3mos for one year and at 5 years
Population: Participants who had data collected for survey. Only participants in group 1 completed survey.
Measure: Number; unit: percentage of participants
Groups:
- Baseline; 1 Month; 3 Months; 6 Month; 9 Months; 12 Months; 5 Years: Patients undergo partial breast irradiation delivered as a single intra-operative radiation dose to the tumor bed.
Arm/Group | Baseline | 1 Month | 3 Months | 6 Month | 9 Months | 12 Months | 5 Years
Number analyzed (Participants) | 12 | 10 | 8 | 5 | 5 | 10 | 6
percentage of participants
  Excellent | 8 | 0 | 13 | 0 | 0 | 10 | 0
  Good | 54 | 50 | 37 | 25 | 20 | 20 | 33
  Fair | 38 | 50 | 37 | 75 | 60 | 60 | 50
  Poor | 0 | 0 | 13 | 0 | 20 | 10 | 17

19. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: Percent of participants indicating total satisfaction or not totally satisfied but would choose same treatment again on QOL survey
  Participants indicate level of satisfaction by answering "my satisfaction about the treatment and results is"
  1. I am totally satisfied with the treatment and results
  2. I am not totally satisfied but would choose the same treatment again.
  3. I am not totally satisfied and would choose the standard 5-6 week course of radiation if I had it to do all over again.
  4. I am dissatisfied with my treatment.
Time Frame: 1 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 12 | 1
percentage of participants | 100 | 100

20. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: as for outcome 19
Time Frame: 3 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 100 | 100

21. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: as for outcome 19
Time Frame: 6 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 100 | 100

22. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: as for outcome 19
Time Frame: 9 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 100 | 100

23. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: as for outcome 19
Time Frame: 12 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 100 | 100

24. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: as for outcome 19
Time Frame: 2 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 100 | 100

25. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: as for outcome 19
Time Frame: 3 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 10 | 1
percentage of participants | 100 | 100

26. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: as for outcome 19
Time Frame: 4 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 10 | 0
percentage of participants | 100 |

27. Primary Outcome: Percent of Participants Indicating Total Satisfaction or Not Totally Satisfied But Would Choose Same Treatment Again on Quality of Life (QOL) Survey
Description: as for outcome 19
Time Frame: 5 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 9 | 0
percentage of participants | 100 |

28. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 1 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 12 | 1
percentage of participants | 33 | 0

29. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 1 month after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 12 | 1
percentage of participants | 8 | 0

30. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 3 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 36 | 0

31. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 6 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 36 | 0

32. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 9 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 36 | 0

33. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 12 month after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 36 | 0

34. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 2 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 36 | 0

35. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 3 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 36 | 0

36. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 4 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 36 | 0

37. Primary Outcome: Percent of Participants Experiencing Complications After Intervention
Description: Overall complication rate, as measured by percent of participants experiencing complications after intervention
Time Frame: 5 years after RT
Population: Evaluable participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 10 | 1
percentage of participants | 40 | 0

38. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 3 month after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

39. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 6 month after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

40. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 9 month after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

41. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 12 month after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

42. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 2 years after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

43. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 3 years after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

44. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 4 years after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 11 | 1
percentage of participants | 9 | 0

45. Secondary Outcome: Percent of Participants With Delayed Wound Healing
Description: Wound healing rate, as measured by percent of participants with delayed wound healing
Time Frame: 5 years after RT
Population: Evaluable participants enrolled on study
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
Number analyzed (Participants) | 10 | 1
percentage of participants | 10 | 0

ADVERSE EVENTS:
Time Frame: up to 5 years
Arm/Group | Intraoperative Radiation Therapy | Intracavitary Balloon Brachytherapy
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/1
Other Adverse Events (participants affected / at risk) | 11/12 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraoperative Radiation Therapy (N=12) | Intracavitary Balloon Brachytherapy (N=1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - nose (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (4) | 0 (0)
Insomnia (General disorders) | 3 (4) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 0 (0)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Breast indentation/dimpling (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin retraction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin dimpling (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 (9) | 1 (2)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Hot flashes/flushes (Endocrine disorders) | 3 (3) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Breast Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Edema: limb (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Edema: trunk/genital (Blood and lymphatic system disorders) | 3 (4) | 1 (2)
Lymphatics: seroma (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibrosis-cosmesis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Superficial soft tissue breast fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Seroma (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (2) | 0 (0)
Mood alteration - Depression (Nervous system disorders) | 2 (3) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0)
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pain - Breast (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain - Dental/teeth/peridontal (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Pain - Head/headache (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Pain - Pelvis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain - Skin (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Breast nipple/areolar deformity (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nipple Inversion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intra-operative injury - Skin (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-05-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT00945061/Prot_SAP_000.pdf